CLINICAL TRIAL: NCT04329793
Title: Effectiveness of a Treatment With the Robot - Assisted Gait Training System Walkbot in Patients With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Raquel Olmos Gómez, Principal investigator, Universidad de Murcia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2365/2019
Record Dates: First submitted 2020-03-07; First posted 2020-04-01 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Assisted gait training with Walkbot System and their usual Physical Therapy.
  Interventions: Device: Assisted gait training with Walkbot System; Other: Physical Therapy
- Control arm (Active Comparator): Their usual Physical Therapy.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Device: Assisted gait training with Walkbot System — The experimental group will receive at least 3 treatment sessions per week consisting of 40 minutes in robot-assisted gait training with Walkbot System in addition to their usual Physical therapy sessions. In total, the number of Walkbot sessions will be 20, in uninterrupted weeks.
  Other Names: Physical Therapy
  Arms: Intervention arm
Other: Physical Therapy — The control group will receive their usual Physical therapy sessions during 6 weeks.

SUMMARY:
The improvement of walking capacity is a key objective of the rehabilitation of children with PC. There are different approaches from physiotherapy to address this need, including walking on the ground and on treadmill with partial weight support. Currently, there are robotic technologies adapted to the functional rehabilitation of patients. Assisted gait training with robotic devices such as the Walkbot allows a longer duration of training, at more variable speeds, and with a constant gait pattern adapted to the patient. This training, based on the intensity and repetition of the movement, has beneficial effects on the recovery and improvement of the patient's postural and locomotor functions.

There are some studies that evaluate walking interventions on treadmill with partial weight support, on the ground and in assisted walking robot in patients with PC.

Currently, there are no studies conducted that report the effectiveness of interventions performed with robotic walking training device Walkbot K on PC. However, studies in adults with Walkbot S, affected with neurological injury, have reported good results.

Assisted gait training with robotic devices such as the Walkbot, based on the intensity and repetition of the movement, has beneficial effects on the recovery and improvement of the patient's postural and locomotor functions. However, due to the little evidence that exists, it is necessary to know the effectiveness of the Walkbot assisted walking robot in these patients by means of a clinical trial that allows to firmly establish the scope of its benefits.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy diagnosis (diplegia or tetraplegia)
* Ability to communicate even if not verbal (yes/not; gestures; pictograms; sounds)
* Levels II, III and IV in GMFCS
* Unsupported seating capacity
* Go on standing with or without help
* Not receiving therapy with a walking robot and not having received it in at least one year

Exclusion Criteria:

* Serious psychiatric problems
* Serious heart problems
* Active tumors
* Severe joint degenerative problems
* Degenerative diseases of the nervous system
* Mitochondrial diseases
* Recent surgeries
* Unbound fractures
* Severe osteoporosis
* Uncontrolled seizures
* Open wounds in the lower half of the body
* Extreme fear of being placed in robotic devices
* Anthropomorphic measures are below the minimum required to use the device

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-03-14 (Actual)

PRIMARY OUTCOMES:
Ability and quality of walking. | Baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention
  Changes in Gross Motor Function Measure-88 (dimensions IV y V)

SECONDARY OUTCOMES:
Functionality and autonomy | Baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention
  Differences in the basic activities of daily life, measured with the PedsQL- Cerebral Palsy Module
Muscle strength | Baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention
  Differences in muscle strength of lower limbs, measured with dynamometer.
Range of motion | Baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention
  Analyze if the range of joint mobility is increased in those joints that are more limited, measured with goniometer.
Spasticity | Baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention
  Changes in spasticity values, measured with the modified Ashworth Scale. Higher scores mean worse outcome. Minimum value is 0. Maximum value is 4.
Quality of walking: Edinburgh Visual Gait Scale | Baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention
  Changes in Edinburgh Visual Gait Scale values. Higher scores mean worse outcome. Minimum value is 0. Maximum value is 34.
Gait endurance | Baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention
  Changes in 6 minutes walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Raquel Olmos Gómez, Yecla, Murcia, Spain

REFERENCES:
- [Derived] Olmos-Gomez R, Calvo-Munoz I, Gomez-Conesa A. Treatment with robot-assisted gait trainer Walkbot along with physiotherapy vs. isolated physiotherapy in children and adolescents with cerebral palsy. Experimental study. BMC Neurol. 2024 Jul 15;24(1):245. doi: 10.1186/s12883-024-03750-9. PMID 39009990